CLINICAL TRIAL: NCT00510237
Title: Intervention Development for Newly Diagnosed Youth With HIV
Brief Title: Intervention for Newly Diagnosed Youth With HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ATN 068
Record Dates: First submitted 2007-07-31; First posted 2007-08-01 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2016-08

CONDITIONS: HIV
Keywords: HIV; Adolescents newly diagnosed with HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): 5-7 females per group at each of the four sites.
  Interventions: Behavioral: "Adolescents Coping, Connecting, Empowering, and Protecting Together" (Project ACCEPT)
- 2 (Experimental): 5-7 males per group at each of the four sites.
  Interventions: Behavioral: "Adolescents Coping, Connecting, Empowering, and Protecting Together" (Project ACCEPT)

INTERVENTIONS:
Behavioral: "Adolescents Coping, Connecting, Empowering, and Protecting Together" (Project ACCEPT) — The intervention will consist of a combination of individual and group-based sessions in which the youth will participate. This combination allows for more intensive individualized attention as well as supportive group sessions. Youth will first participate in two individual sessions, followed by nine group sessions, and end with one additional individual session.

SUMMARY:
This study will pilot test an HIV intervention for newly diagnosed youth (diagnosed for less than 15 months) to assess its acceptability and feasibility preliminary to and leading up to a full-scale, randomized trial. The general focus of the intervention is to aid in the psychosocial adjustment of adolescents who have recently been diagnosed with HIV.

DETAILED DESCRIPTION:
The intervention will consist of a combination of individual and group-based sessions in which the youth will participate. This combination allows for more intensive individualized attention as well as supportive group sessions. Youth will first participate in two individual sessions, followed by nine group sessions, and end with one additional individual session.

Individual Session I: Orientation I

Part A - meet with interventionist for ecological assessment, rapport building, and preparation for meeting with medical provider Part B - meet with medical provider to answer HIV specific medical questions (i.e., transmission information, viral load/t-cells, opportunistic infections,etc.). The interventionist will be present in Part B as well.

Individual Session II: Orientation II

Part A - meet with interventionist for continued debriefing, question/answer, preparation for group participation.

Part B - meet with peer facilitator to discuss individual experiences living with HIV, rapport building, peer-specific questions. The interventionist will be present in Part B as well.

Individual session III: Wrap-up and Action Planning (to take place after group sessions are complete)

Part A - action plan with linkage to identified agencies via facilitated referrals Part B - (optional) support building - participants may bring parents, partner, friend, or other potential source of support for question/answer session with interventionist

Session I: Developing Group Cohesion

- Icebreaker, team building, group rules, facilitation of group "ownership" by participants.

Session II: Disclosure, Stigma & Relationships

* Disclosure to family, friends, peers and co-workers as well as dealing with stigma associated with HIV/AIDS;
* Concerns about current or future romantic and/or sexual relationships, including discussion of safer sex, condom use, sero-discordant couples.

Session III: Preparing for Medical Intervention

- Working with medical providers, an overview of clinic appointments and expectations surrounding attendance, a preliminary discussion of medications, side effects, and medical management as well as strategies for adherence.

Session IV: Healthy Living

* Issues related to drugs and alcohol;
* Leisure activities such as sports and entertainment;
* Self-care including nutrition and exercise;
* The importance of school and work.

Session V: Stress Reduction/Relaxation & Spirituality

* Techniques including deep breathing, progressive muscle relaxation, visualization, meditation and self-hypnosis;
* Self-care including complimentary therapies such as massage and acupuncture
* Spirituality;
* Planning social outings and activities.

Session VI: Gender Specific

* Males: issues surrounding sexuality and sexual orientation, male role of caring for self, loved ones, and the community;
* Females: issues surrounding sexuality, pregnancy and parenting, female role of caring for self, loved ones, and the community.

Session VII: Self-Esteem/Self-Worth

- Strategies to improve self-esteem and self-worth;

Session VIII: Legal Issues/Advocacy

* Legal rights and advocacy;
* Linkage to community advocacy groups;
* Preparing to become a speaker/advocate;
* Health insurance/life insurance.

Session IX: Future Planning

- Planning for the future including issues related to work and school (e.g., job application process, applying for financial aid), job training and career choices.

ELIGIBILITY:
Inclusion Criteria:

To be considered eligible for enrollment in ATN 068, a participant must meet the criteria listed below:

* Receive services at one of the 4 selected ATN sites or their community partners;
* HIV-infected as documented by medical record review or verbal verification with referring professional;
* Received HIV diagnosis less than 15 months ago as documented by medical record review or verbal verification with referring professional;
* Fall between the ages of 16-24 (inclusive) at the time of informed consent/assent;
* Must be willing to participate in the both the individual and group sessions;
* Give informed consent/assent for study participation.

Exclusion Criteria:

Participants who meet any of the exclusion criteria listed below are considered ineligible:

* Acquired HIV through perinatal infection;
* Presence of serious psychiatric symptoms (active hallucinations, thought disorder);
* Visibly distraught (suicidal, homicidal, exhibiting violent behavior);
* Intoxicated or under the influence of alcohol or other substances at the time of study enrollment.

Ages: 16 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2007-02; Primary Completion 2008-06 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
The best procedures for a larger trial (e.g. timing, content etc. of ACASI administration) | 7 months
The appropriateness of specific instruments proposed. | 7 months
The perceived sensitivity of measures to change over time. | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Sybil Hosek, PhD, Study Chair — John Stroger Jr. Hospital of Cook County
Locations (4):
- United States (4):
  - University of Miami School of Medicine, Miami, Florida
  - John Stroger Jr. Hospital of Cook County, Chicago, Illinois
  - Montefiore Medical Center, The Bronx, New York
  - St. Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- See also: Website for the Adolescents Trials Network for HIV/AIDS Interventions — http://www.atnonline.org